CLINICAL TRIAL: NCT01864408
Title: Interactive Patient and Provider Counseling on Pelvic Organ Prolapse: Do Patients Better Understand and Do Providers Better Counsel
Brief Title: Interactive Web-Based Tool for Pelvic Organ Prolapse: Impact on Patient Understanding and Provider Counseling
Acronym: iPad
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 12-0332
Record Dates: First submitted 2013-05-13; First posted 2013-05-29 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2013-05

CONDITIONS: Pelvic Organ Prolapse
Keywords: Patient counseling; Patient satisfaction; Pelvic organ prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse; Patient Satisfaction | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Other): Group 1: subjects will receive "usual practice" counseling regarding pelvic organ prolapse after new patient history and physical exam.
  Interventions: Other: "Usual practice" counseling
- Group 2 (Experimental): Group 2: subjects will receive "usual practice" counseling in addition to interactive patient/provider counseling using the pelvic organ prolapse web-based tool (iPad) after new patient history and physical exam.
  Interventions: Other: Standard "usual practice" clinical counseling with the pelvic organ prolapse web-based tool (iPad).

INTERVENTIONS:
Other: "Usual practice" counseling
  Other Names: Standard "usual practice" clinical counseling routinely performed after new patient history and physical exam.
  Arms: Group 1
Other: Standard "usual practice" clinical counseling with the pelvic organ prolapse web-based tool (iPad). — After a new patient history and physical exam, with POP-Q exam, the subjects specific exam findings are entered into the Interactive Pelvic Organ Prolapse Quantification (POP-Q) Program. The program then constructs a cartoon of the subjects physical exam findings. This image is then used in counseling in addition to standard "usual practice" counseling.
  Other Names: Interactive Pelvic Organ Prolapse Quantification (POP-Q) Program.
  Arms: Group 2

SUMMARY:
The primary aim is to assess whether an interactive patient/provider counseling process using a web-based tool (iPadTM) will improve patient satisfaction regarding understanding of her bulge symptoms.

The secondary aims are to assess whether an interactive patient/provider counseling process using web-based tool (iPadTM) will:

1. Decrease patient anxiety with counseling
2. Improve patient satisfaction with counseling
3. Improve provider knowledge, anxiety, and satisfaction with counseling
4. Be easy to use in clinic
5. Be actually used in clinic

DETAILED DESCRIPTION:
This will be a randomized controlled trial comparing conventional counseling regarding pelvic organ prolapse versus an interactive patient/provider counseling process using a pelvic organ prolapse web-based tool (iPad).

All women agreeing to enroll will:

1. Complete a pre-visit questionnaire querying

   1. Baseline satisfaction with knowledge of their presenting bulge symptoms ("pelvic anatomy")
   2. Anxiety related to their presenting symptoms
2. Undergo a new patient history and physical exam, including a pelvic organ prolapse quantification (POPQ) exam as per practice standard.
3. Patients will then be randomized and will either receive:

   1. Group 1: "usual practice" counseling regarding pelvic organ prolapse
   2. Group 2: "usual practice" counseling in addition to interactive patient/provider counseling using the pelvic organ prolapse web-based tool (iPad)
4. Complete a post-visit questionnaire before leaving the office querying:

   1. Post-visit satisfaction with knowledge of their presenting bulge symptoms ("pelvic anatomy")
   2. Anxiety related to their presenting symptoms
   3. Satisfaction with counseling received regarding their presenting bulging symptoms.

Provider assessment:

The providers participating in this study will:

1. Complete a pre-trial questionnaire assessing satisfaction with knowledge and anxiety regarding counseling, and satisfaction with ability to counsel women regarding pelvic organ prolapse.
2. Watch a 2 minute video tutorial educating them on the use of the web-based interactive tool
3. Complete a post-trial questionnaire assessing satisfaction with knowledge and anxiety regarding counseling, and satisfaction with ability to counsel women regarding pelvic organ prolapse.

Powering the Study:

Assuming a 30% difference in satisfaction with knowledge of presenting bulge symptoms/ "pelvic anatomy", this study will enroll 45 pts in each arm (total of 90 pts) to achieve a power of 80% and an alpha of 0.05.

Analytic Plan: Statistical analysis will be performed with SPSS v 19.0 (Chicago, IL) and will include, where appropriate, categorical data analysis (Pearson chi-square, Fisher's Exact),continuous data analysis (Student's t-test, Mann-Whitney-U), and Pearson correlation, and logistic regression analyses where appropriate.

DATA COLLECTION:

Data will be collected by the project personnel. Patient demographic and physical exam data will be collected by physician members of the project personnel team during the single patient-visit of this trial. The physician members of the project personnel team will perform either the "usual practice" or "usual practice" plus "interactive, web-based tool-facilitated" patient counseling. Patient and provider questionnaire data will also be collected by the project personnel team.

Number and duration of subject contact: All data will be collected over the course of a patient's single "New Patient" visit. There will be no patient follow-up after this single visit.

ELIGIBILITY:
Inclusion Criteria:

Patients

* English speaking
* Women over the age of 18
* With complaints of symptomatic bulging from the vagina
* Presenting as a new patient to University of North Carolina, Chapel Hill (UNC) Urogynecology clinic

Providers

* All providers at UNC Urogynecology clinic will be allowed to participate in counseling sessions

Exclusion Criteria:

* Patients not meeting inclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in patient reported satisfaction with understanding of bulge symptoms based on Likert scale scores. | Day 1
  Immediately before a history, physical, and counseling session subjects will fill out a Likert scale questionnaire (1=Very Dissatisfied, 2=Dissatisfied, 3=Neutral, 4=Satisfied, 5=Extremely Satisfied) to evaluate pre-visit satisfaction with understanding of bulge symptoms. After the history and physical exam subjects are randomized to group 1 or 2 for their counseling session. After the counseling session, they will fill out a similar Likert scale questionnaire to assess their satisfaction with understanding of their bulge symptoms. We will then compare the pre-visit and post-visit satisfaction with understanding of bulge symptoms for each group.

SECONDARY OUTCOMES:
Change in patient reported anxiety with understanding of bulge symptoms based on Likert scale scores. | Day 1
  Immediately before a history, physical, and counseling session subjects will fill out a Likert scale questionnaire (1=Not at all Anxious, 2=A little Anxious, 3=Moderately Anxious, 4=Very Anxious, 5=Extremely Anxious) to evaluate pre-visit anxiety related to bulge symptoms. After the history and physical exam subjects are randomized to group 1 or 2 for their counseling session. After the counseling session, they will fill out a similar Likert scale questionnaire to assess their anxiety regarding their bulge symptoms. We will then compare the pre-visit and post-visit anxiety related to bulge symptoms for each group.
Assessment of patient satisfaction after standard counseling (group 1) vs standard counseling with a web-based tool (ipad)(group 2). | Day 1
  At the end of the visit, Subjects will fill out a Likert scale questionnaire to evaluate overall satisfaction (1=Very Dissatisfied, 2=Dissatisfied, 3=Neutral, 4=Satisfied, 5=Extremely Satisfied) with counseling method received.
Change in provider satisfaction with knowledge and anxiety regarding counseling and satisfaction with the ability to counsel women regarding pelvic organ prolapse. | Baseline and at 9 months
  All providers will fill out a Likert scale questionnaire to evaluate pre-study satisfaction with knowledge and anxiety regarding counseling and satisfaction with the ability to counsel women regarding pelvic organ prolapse. They will again complete the a similar questionnaire at the end of the study.
Provider assessment: was the web-based tool easy to use, would you implement this tool into your practice? | At 9 months
  All providers will fill out a Likert scale questionnaire regarding iPad ease of use. They will also be asked if they planned to implement this tool into their practice (Y/N).

CONTACTS AND LOCATIONS:
Overall Officials: Erinn M Myers, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States